CLINICAL TRIAL: NCT05272878
Title: Impact of a Treatment With Angiotensin Receptor Blocker on Outcome After Acute Kidney Injury in Patients Discharged From the ICU "START-or-NOT Trial". A Prospective, Randomized, Double Blinded, Multicenter Study
Brief Title: Impact of a Treatment With Angiotensin Receptor Blocker on Outcome After Acute Kidney Injury in Patients Discharged From the ICU.
Acronym: START-or-NOT
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: APHP200040
Record Dates: First submitted 2022-01-10; First posted 2022-03-10 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-06

CONDITIONS: Acute Kidney Injury
Keywords: Angiotensin-Converting-Enzyme Inhibitor; angiotensin-receptor blockers
MeSH Terms: conditions — Acute Kidney Injury | interventions — Irbesartan; Tablets

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Treatments will be conditioned and labelled by the Contract manufacturing organization AGEPS according to a list provided by an independent person and assigning a treatment arm to each treatment number.
  Randomization and treatment numbers lists are kept strictly confidential until the time of unblinding, and will not be accessible by anyone involved in the study, with the exception of the independent, unblinded statistician approving the randomization scheme; the study will be kept blinded to patients, investigators and study personnel also during the entire study period; The identification of treatment will be concealed by the use of a matching placebo to the study product that will be provided in boxes identical in packaging, labeling and appearance
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- IRBESARTAN (Active Comparator): IRBESARTAN will be introduced at 150 mg orally one daily, with a progressive increase to 300 mg a day, at 7 days or 2 months follow-up visit, based on clinical and biological tolerance. Treatment will be continued for 12 months, unless a side effect would occur.
  Interventions: Drug: IRBESARTAN, tablet, 150 mg
- Placebo (Placebo Comparator): Placebo will be introduced at 150 mg orally one daily, with a progressive increase to 300 mg a day, at 7 days or 2 months follow-up visit, based on clinical and biological tolerance. Treatment will be continued for 12 months, unless a side effect would occur.
  Interventions: Drug: Placebo, tablet, 150 mg

INTERVENTIONS:
Drug: IRBESARTAN, tablet, 150 mg — IRBESARTAN will be introduced at 150 mg orally one daily, with a progressive increase to 300 mg a day, at 7 days or 2 months follow-up visit.Treatment will be continued for 12 months, unless a side effect would occur.
  Arms: IRBESARTAN
Drug: Placebo, tablet, 150 mg — Placebo will be introduced at 150 mg orally one daily, with a progressive increase to 300 mg a day, at 7 days or 2 months follow-up visit.Treatment will be continued for 12 months, unless a side effect would occur.
  Arms: Placebo

SUMMARY:
The patients discharged from intensive care units (ICU) have a high incidence of cardiovascular events and mortality rate during the year following ICU discharge. Among patients admitted to the ICU, patients with acute kidney injury (AKI) display high risk of such events. The investigators furthermore demonstrated that AKI could induce remote cardio-vascular injury and fibrosis, which may be involved in the poor prognosis of AKI. Strategies that may prevent the cardiovascular consequences of AKI in most severe patients (i.e. post-AKI ICU survivors) may therefore improve long term outcomes.

AKI has been associated with activation of the renin-angiotensin-aldosterone system (RAAS). Activation of the RAAS has been further associated with long-term health consequences especially with cardiovascular damages. Potential protective effects of RAASi following acute injury have been reported in observational studies. With this randomized controlled trial, the investigators aim at investigating the impact of treatment with RAAS inhibitors after AKI on cardiovascular and kidney outcomes.

DETAILED DESCRIPTION:
Phase III study Prospective, multicenter, superiority, double-blind, randomized controlled study with two arms (1:1).

* Inclusion of patients who are discharged alive (or ready to be discharged) from ICU or acute care and developed acute kidney injury during the ICU stay (according to the KDIGO criteria) - and signing of the consent to participate at this research
* Enrolled patients will be randomly assigned to one of the two study groups once their renal function has stabilized for at least 48 hours and within 30 days from ICU or acute care discharge. Patients randomized will be stratified according to the center and the severity of AKI during ICU stay (KDIGO 1 vs KDIGO 2 or 3)
* All patients with have a clinical examination and biological visit (i.e. serum creatinine, potassium, and NT-ProBNP) 7(+/-2) days after inclusion, at 2 months, 6 months and at 12 months. Microalbuminuria will be further measure at inclusion and 12 months. In the control and treatment group, treatment will be upgraded to 2 pills (IRBESARTAN 150 mg or Placebo) if Serum creatinine has not risen by more than 30% since previous visit and no hyperkalemia and no hypotension are noticed. Treatment management will be performed by intensivists, nephrologists or cardiologists involved in the protocol.

Biological collection

A plasma and urine collected as part of the study will be stored in a biological sample collection at inclusion and at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Patient between 18 and 75 years old
* Met criteria for acute kidney injury during the ICU stay (according to the KDIGO criteria)
* After their renal function has stabilized for at least 48 hours (Serum creatinine decreasing or not increasing more than 26 micromol/L or 25%) among patients ready to be discharged from the ICU or acute careTCU. and within 30 days after their ICU discharge.
* Signed informed consent
* Patients affiliated to a Social Security System
* Women of childbearing potential and men must agree, to use adequate and highly effective contraception, until the end of the research.

Exclusion Criteria:

* Patient treated with ACEi or ARB before ICU admission
* Patient for whom treatment with ACEi or ARB is strongly recommended according to the international guidelines at discharge (i.e. patients with congestive heart failure and persistent dyspnea with LVEF<40%,, patients with diabetes mellitus and either albuminuria > 300 µg/g creatininuria or hypertension associated with microalbuminuria or hypertension associated with eGFR < 60 ml/min) known before ICU admission.
* Hyperkalemia>5 mmol/L
* Systolic blood pressure <100 mmHg
* Patient with severe renal failure, as defined by estimated glomerular filtration rate creatinine clearance < 15 ml/min/1.73m2), requiring renal replacement therapy at ICU discharge
* Oral route impossible.
* Pregnancy
* Breast feeding
* Patients chronically treated with Aliskiren
* Known hypersensitivity to the active substance or to one of its excipients and in particular to lactose
* Patients with known primary hyperaldosteronism
* Patients with known severe and symptomatic aortic stenosis, mitral stenosis or obstructive hypertrophic cardiomyopathy.
* Patients treated with lithium
* Patient undergoing psychiatric care
* Inability to consent due to psychiatric disorders defined as psychiatric disorders or patient with a mental state requiring immediate care with either by constant medical surveillance justifying hospitalization, or regular medical follow-up justifying specific treatment
* Patient deprived of liberty by a judicial or administrative decision
* Patient to a legal protection measure (guardianship, curatorship and safeguard of justice)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 508 (Estimated)
Dates: Start 2022-11-22 (Actual); Primary Completion 2025-06-27 (Actual); Study Completion 2026-06-27 (Estimated)

PRIMARY OUTCOMES:
Time to MACE (major adverse cardiovascular events) | Within the year after randomization
  cardiovascular events will be defined as: acute heart failure, stroke, acute coronary syndrome

SECONDARY OUTCOMES:
Occurrence of chronic kidney disease | one year after ICU discharge
  kidney disease defined as eGFR <60 ml/min/1.73m2
Albuminuria>0.3 g/day one year after ICU discharge | one year after ICU discharge
Chronic kidney disease staging | One year after randomization
Change in Chronic kidney disease staging | One year after randomization
New episode of acute kidney injury requiring hospitalization | within one year after randomization
  Acute kidney injury according to the KDIGO criteria
Hyperkalemia >6 mmol/L | within one year after randomization
Death | within one year after randomization

CONTACTS AND LOCATIONS:
Overall Officials: Etienne Gayat, MD-PhD, Principal Investigator — APHP-Hôpital Lariboisière; Matthieu Legrand, MD-PhD, Study Director — Departement of Anesthesia and Peri-operative Care, UCSF
Locations (1):
- Hospital Lariboisière, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Grams ME, Rabb H. The distant organ effects of acute kidney injury. Kidney Int. 2012 May;81(10):942-948. doi: 10.1038/ki.2011.241. Epub 2011 Aug 3. PMID 21814177
- [Background] Burchill L, Velkoska E, Dean RG, Lew RA, Smith AI, Levidiotis V, Burrell LM. Acute kidney injury in the rat causes cardiac remodelling and increases angiotensin-converting enzyme 2 expression. Exp Physiol. 2008 May;93(5):622-30. doi: 10.1113/expphysiol.2007.040386. Epub 2008 Jan 25. PMID 18223026
- [Background] Chou YH, Huang TM, Pan SY, Chang CH, Lai CF, Wu VC, Wu MS, Wu KD, Chu TS, Lin SL. Renin-Angiotensin System Inhibitor is Associated with Lower Risk of Ensuing Chronic Kidney Disease after Functional Recovery from Acute Kidney Injury. Sci Rep. 2017 Apr 13;7:46518. doi: 10.1038/srep46518. PMID 28406186
- [Background] Gayat E, Hollinger A, Cariou A, Deye N, Vieillard-Baron A, Jaber S, Chousterman BG, Lu Q, Laterre PF, Monnet X, Darmon M, Leone M, Guidet B, Sonneville R, Lefrant JY, Fournier MC, Resche-Rigon M, Mebazaa A, Legrand M; FROG-ICU investigators. Impact of angiotensin-converting enzyme inhibitors or receptor blockers on post-ICU discharge outcome in patients with acute kidney injury. Intensive Care Med. 2018 May;44(5):598-605. doi: 10.1007/s00134-018-5160-6. Epub 2018 May 15. PMID 29766216
- [Background] Brar S, Ye F, James MT, Hemmelgarn B, Klarenbach S, Pannu N; Interdisciplinary Chronic Disease Collaboration. Association of Angiotensin-Converting Enzyme Inhibitor or Angiotensin Receptor Blocker Use With Outcomes After Acute Kidney Injury. JAMA Intern Med. 2018 Dec 1;178(12):1681-1690. doi: 10.1001/jamainternmed.2018.4749. PMID 30422153
- [Background] Wang HE, Muntner P, Chertow GM, Warnock DG. Acute kidney injury and mortality in hospitalized patients. Am J Nephrol. 2012;35(4):349-55. doi: 10.1159/000337487. Epub 2012 Apr 2. PMID 22473149
- [Background] Go AS, Hsu CY, Yang J, Tan TC, Zheng S, Ordonez JD, Liu KD. Acute Kidney Injury and Risk of Heart Failure and Atherosclerotic Events. Clin J Am Soc Nephrol. 2018 Jun 7;13(6):833-841. doi: 10.2215/CJN.12591117. Epub 2018 May 17. PMID 29773712
- [Background] Lee BJ, Hsu CY, Parikh RV, Leong TK, Tan TC, Walia S, Liu KD, Hsu RK, Go AS. Non-recovery from dialysis-requiring acute kidney injury and short-term mortality and cardiovascular risk: a cohort study. BMC Nephrol. 2018 Jun 11;19(1):134. doi: 10.1186/s12882-018-0924-3. PMID 29890946
- [Background] Omotoso BA, Abdel-Rahman EM, Xin W, Ma JZ, Scully KW, Arogundade FA, Balogun RA. Dialysis requirement, long-term major adverse cardiovascular events (MACE) and all-cause mortality in hospital acquired acute kidney injury (AKI): a propensity-matched cohort study. J Nephrol. 2016 Dec;29(6):847-855. doi: 10.1007/s40620-016-0321-6. Epub 2016 Jun 15. PMID 27307250
- [Background] Bansal N, Matheny ME, Greevy RA Jr, Eden SK, Perkins AM, Parr SK, Fly J, Abdel-Kader K, Himmelfarb J, Hung AM, Speroff T, Ikizler TA, Siew ED. Acute Kidney Injury and Risk of Incident Heart Failure Among US Veterans. Am J Kidney Dis. 2018 Feb;71(2):236-245. doi: 10.1053/j.ajkd.2017.08.027. Epub 2017 Nov 20. PMID 29162339